CLINICAL TRIAL: NCT07086326
Title: A Prospective, Randomized, Open-label, Controlled Phase Ⅱ Clinical Trial of Ivonescimab Combined With Chemotherapy Versus Penpulimab Combined With Chemotherapy for Neoadjuvant Treatment of Non-small Cell Lung Cancer (NSCLC)
Brief Title: A Phase II Randomized Trial of Neoadjuvant Ivonescimab or Penpulimab Plus Chemotherapy in Resectable NSCLC
Acronym: NEOINSPIRE
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Yang Fan, MD (Other)
Responsible Party: Sponsor-Investigator, Yang Fan, MD, Peking University People's Hospital, Peking University People's Hospital
Organization: Peking University People's Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AK112-IIT-014
Record Dates: First submitted 2025-07-17; First posted 2025-07-25 (Actual); Last update posted 2025-07-25 (Actual); Status verified 2025-07

CONDITIONS: NSCLC; Neoadjuvant Therapy; Immunotherapy; AK112; Bispecific Antibody

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Ivonescimab+Chemo (Experimental): Ivonescimab (AK112) + platinum-based doublet chemotherapy as neoadjuvant treatment, administered every 3 weeks (Q3W) for 3-4 cycles. Surgical resection should be performed 4-6 weeks after the last dose, followed by safety follow-up and survival surveillance.
  Interventions: Drug: Ivonescimab+Chemo
- Penpulimab+Chemo (Active Comparator): Penpulimab (AK105) + platinum-based doublet chemotherapy as neoadjuvant treatment, administered every 3 weeks (Q3W) for 3-4 cycles. Surgical resection should be performed 4-6 weeks after the last dose, followed by safety follow-up and survival surveillance.
  Interventions: Drug: Penpulimab+Chemo

INTERVENTIONS:
Drug: Ivonescimab+Chemo — Ivonescimab (AK112) + platinum-based doublet chemotherapy
  Arms: Ivonescimab+Chemo
Drug: Penpulimab+Chemo — Penpulimab (AK105) + platinum-based doublet chemotherapy
  Arms: Penpulimab+Chemo

SUMMARY:
This is a randomized, open-label, multicenter phase II study. The trial plans to enroll 164 subjects with resectable stage IIA-IIIB (N2) NSCLC. Participants will be randomized 1:1 into either the ivonescimab plus chemotherapy or penpulimab plus chemotherapy treatment arm. After 3-4 cycles of neoadjuvant therapy, surgical resection will be performed. The primary objective is to compare the pathological complete response (pCR) rate assessed by local pathologists between ivonescimab-based and penpulimab-based chemo-immunotherapy regimens in the neoadjuvant treatment of resectable NSCLC.

ELIGIBILITY:
Inclusion Criteria:

1. Voluntarily sign the written Informed Consent Form (ICF) and consent to receive curative surgical treatment.
2. Participants must be aged ≥ 18 years, regardless of gender.
3. Eastern Cooperative Oncology Group (ECOG) Performance Status Score is 0-1.
4. Histologically confirmed resectable Stage IIA-IIIB (N2) non-small cell lung cancer (NSCLC) according to the 9th edition of the TNM staging system for lung cancer by the Union for International Cancer Control (UICC) and the American Joint Committee on Cancer (AJCC).
5. Prior to study enrollment, subjects must be evaluated by an attending thoracic surgeon responsible for the surgery to verify eligibility for R0 resection with curative intent.
6. NSCLC appears solid or subsolid (not purely ground-glass opacity [GGO]) on CT scan. For subsolid lesions, tumor size (i.e., clinical T stage) should be based solely on the solid component without measuring the GGO portion.
7. Normal pulmonary function test results.
8. At least one measurable lesion according to RECIST v1.1, amenable to repeated accurate measurements.
9. Adequate cardiac function.
10. Laboratory values obtained during screening or within ≤14 days prior to randomization indicate adequate organ function.
11. For patients planned to receive cisplatin: No hearing impairment.
12. Women of childbearing potential must have a negative pregnancy test result within 3 days before first treatment; all subjects (male and female) must agree to use appropriate contraceptive methods during the study.

Exclusion Criteria:

1. Patients with large cell neuroendocrine carcinoma (LCNEC) or NSCLC mixed with small cell lung cancer components;
2. Presence of locally advanced unresectable disease (any stage) or metastatic disease (Stage IV). Subjects with contralateral mediastinal lymph node involvement confirmed by PET-CT scan.
3. NSCLC diagnosed with EGFR-sensitive mutations or ALK gene translocation. For non-squamous cell carcinoma subjects (including NSCLC with unclear pathology), tumor tissue-based EGFR and ALK testing results must be provided. If EGFR/ALK status is unknown, testing must be performed prior to enrollment. For squamous NSCLC subjects, EGFR/ALK testing is not required during screening if status is unknown.
4. Any prior systemic or local anti-tumor therapy for NSCLC;
5. Concurrent enrollment in another clinical trial;
6. History of other malignancies (excluding NSCLC) within 3 years prior to randomization;
7. Active autoimmune disease requiring systemic treatment within 2 years prior to randomization;
8. History of major diseases within 1 year prior to randomization;
9. Severe cardiovascular risk factors;
10. History of significant bleeding diathesis or coagulation disorders; clinically significant bleeding symptoms (including but not limited to gastrointestinal hemorrhage, hemoptysis ≥1 teaspoon of fresh blood/clots or pure hemoptysis without sputum, minor blood-tinged sputum allowed; excluding epistaxis and retracted blood-tinged nasal discharge) within 4 weeks prior to randomization;
11. Any other conditions deemed unsuitable for enrollment by the investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 164 (Estimated)
Dates: Start 2025-07-31 (Estimated); Primary Completion 2026-12-30 (Estimated); Study Completion 2027-12-30 (Estimated)

PRIMARY OUTCOMES:
Pathologic Complete Response (pCR) Rate | Within 1 month after surgery
  Pathologic complete response (pCR) rate is defined as the percentage of participants with no residual viable tumor in lung primary or lymph nodes as evaluated by systematic pathological review of surgical specimens.

SECONDARY OUTCOMES:
Major Pathologic Response (MPR) Rate | Within 1 month after surgery
  Major pathologic response (MPR) rate is defined as the percentage of participants with less than 10% of residual viable tumor in lung primary or lymph nodes as evaluated by systematic pathological review of surgical specimens. Viable tumors in situ carcinoma should not be included in MPR calculation.
Event-Free Survival (EFS) | the time from the first dose to the occurrence of any of the following events (whichever occurs first), assessed in the Intention-To-Treat (ITT) population: Disease progression (based on RECIST v1.1 criteria by investigators); Local recurrence or dist
  Defined as the time from the first dose to the occurrence of any of the following events (whichever occurs first), assessed in the Intention-To-Treat (ITT) population: Disease progression (based on RECIST v1.1 criteria by investigators); Local recurrence or distant metastasis; Death from any cause

OTHER OUTCOMES:
Deep pathologic response (DPR) rate | Within 1 month after surgery
  Deep pathologic response (DPR) rate is defined as the percentage of participants with less than 5% of residual viable tumor in lung primary or lymph nodes as evaluated by systematic pathological review of surgical specimens. Viable tumors in situ carcinoma should not be included in DPR calculation.
Objective response rate（ORR） | Within 1 month after surgery
  Preoperative radiological evaluation (as assessed by the investigator according to RECIST v1.1) of the number of complete or partial responses as a proportion of the population in the cohort.
Overall Survival (OS) | The time from the date of randomization to the date of death due to any cause
  Defined as the time from the date of randomization to the date of death due to any cause in the Intention-To-Treat (ITT) population.
2-Year/3-year EFS rate | At 2 and 3 years after randomization
  Defined as the proportion of patients without EFS events at 2 and 3 years after randomization estimated using the Kaplan-Meier method
Incidence of Adverse Events | up to 1 month post surgery
  AE captured by CTCAE 5.0

CONTACTS AND LOCATIONS:
Locations (5):
- China (5):
  - Peking University People's Hospital, Beijing, Beijing Municipality
  - Hunan Cancer Hospital, Changsha, Hunan
  - Shanghai Chest Hospital, Shanghai, Shanghai Municipality
  - The First Affiliated Hospital of Xi'an Jiaotong University, Xi’an, Shanxi
  - Second Affiliated Hospital, School of Medicine, Zhejiang University, Hangzhou, Zhejiang

IPD SHARING:
Plan to Share IPD: No